CLINICAL TRIAL: NCT05405608
Title: The Effect of Intravenous Ondansetron on Reducing Hypotension Due to Bone Cement Syndrome in Total Knee Prosthesis Surgery
Brief Title: The Effect of iv Ondansetron on Reducing Hypotension Due to BCIS in Total Knee Prosthesis Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Prof. Dr., Ataturk University
Other Study IDs: B.30.2.ATA.0.01.00/372
Record Dates: First submitted 2022-05-23; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Bone Cement Syndrome
Keywords: Bone cement syndrome; Hypotension; Ondansetron
MeSH Terms: conditions — Hypotension | interventions — Ondansetron

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group O: Ondansetron applied only, no tourniquet applied
  Interventions: Drug: Ondansetron
- Group TO: Ondansetron and tourniquet applied,
  Interventions: Drug: Ondansetron
- Group S: No ondansetron and tourniquet applied
- Group TS: Ondansetron not applied, only tourniquet applied

INTERVENTIONS:
Drug: Ondansetron — hemodynamic stability in orthopedic surgeries
  Groups: Group O; Group TO

SUMMARY:
Bone cement implantation syndrome (BCIS) is a complication associated with the implantation of polymethylmethacrylate bone cement. Hypoxia, hypotension, and/or unexpected loss of consciousness often result from cementation, prosthetic placement, joint reduction, or tourniquet removal; It is a major cause of intraoperative and postoperative morbidity and mortality. Therefore, reducing the occurrence and severity of BCIS is an important issue.

BCIS is mainly known for its association with hip hemiarthroplasty, total hip arthroplasty (TKA), and vertebroplasty, but is also seen during total knee arthroplasty (TKA). The incidence and associated mortality of BCIS has been investigated only in cemented hemiarthroplasty after displaced femoral neck fractures and in operations performed with cemented TCA and hemiarthroplasty in cancer patients.

To our knowledge, the incidence associated with BCIS (compared to hemiarthroplasty or TKA), associated factors, and mortality for other hips, knee, or shoulder arthroplasty is not yet known. Little is known about the incidence, mortality risk, and factors associated with the development of BCIS during hip hemiarthroplasty and cemented arthroplasty procedures other than primary TKA.

The pathophysiology of BCIS is unclear. The first theories focused on circulating MMA monomers; however, recent evidence suggests an embolism-mediated model. Other additional theories focus on the role of histamine release, complement activation, and finally the multimodal possibilities of all these factors together.

Ondansetron, a 5-hydroxytryptamine 3 (5-HT3) receptor antagonist, has been given preoperatively and intraoperatively to block serotonin-induced pulmonary vasoconstriction.

This study aimed to investigate whether blocking type 3 serotonin receptors with intravenous ondansetron would reduce hypotension due to bone cement syndrome in patients undergoing TKA under combined spinal-epidural anesthesia.

DETAILED DESCRIPTION:
THE EFFECT OF INTRAVENOUS ONDANSETRON ON REDUCING HYPOTENSION DUE TO BONE CEMENT SYNDROME IN TOTAL KNEE PROSTHESIS SURGERY: A RANDOMIZED CONTROLLED THREE-BLIND STUDY

Bone cement implantation syndrome (BCIS) is a complication associated with the implantation of polymethylmethacrylate bone cement. Hypoxia, hypotension, and/or unexpected loss of consciousness often result from cementation, prosthetic placement, joint reduction, or tourniquet removal; It is a major cause of intraoperative and postoperative morbidity and mortality (1). Therefore, reducing the occurrence and severity of BCIS is an important issue.

Donaldson et al.; developed a classification system for BCIS severity. Grade 0: no hypotension/hypoxia, Grade 1: moderate hypoxia (SpO2 <94%) or hypotension [> 20% decrease in systolic blood pressure (SBP) from baseline], Grade 2: severe hypoxia (SpO2 <88%) or hypotension (SBP> 40% decrease in systolic blood pressure (SBP) from baseline) or unexpected loss of consciousness, Grade 3: cardiovascular collapse requiring cardiopulmonary resuscitation (1).

BCIS is mainly known for its association with hip hemiarthroplasty, total hip arthroplasty (TKA), and vertebroplasty, but is also seen during total knee arthroplasty (TKA). The incidence and associated mortality of BCIS has been investigated only in cemented hemiarthroplasty after displaced femoral neck fractures and in operations performed with cemented TCA and hemiarthroplasty in cancer patients (2,3). To our knowledge, the incidence associated with BCIS (compared to hemiarthroplasty or TKA), associated factors, and mortality for other hips, knee, or shoulder arthroplasty is not yet known. Little is known about the incidence, mortality risk, and factors associated with the development of BCIS during hip hemiarthroplasty and cemented arthroplasty procedures other than primary TKA. Rachid Rassir MD et al.; found that 26% of patients developed BCIS after arthroplasty and 6% of all patients experienced severe BCIS (4).

Severe BCIS (Grades 2 and 3) is more common in patients undergoing hip hemiarthroplasty and hip-knee revision arthroplasty, while less common in patients undergoing unicondylar knee arthroplasty and shoulder arthroplasty (4). The pathophysiology of BCIS is unclear. The first theories focused on circulating MMA monomers; however, recent evidence suggests an embolism-mediated model (1,5). Other additional theories focus on the role of histamine release, complement activation, and finally the multimodal possibilities of all these factors together (1,5). The origin of the embolism may be fat, bone marrow, cement, air, bone, or platelet aggregates. Embolism travels to the lungs, heart, and cerebral and coronary circulations (1,5,6). The main clinical problem is acute right ventricular failure due to pulmonary embolism. In addition, bone cement embolism can mechanically induce endothelial injury, which produces reflex vasoconstriction through the release of endothelial mediators. Embolic agents also directly increase PVR by increasing blood thrombin and tissue thromboplastin levels. It can cause a decrease in systemic vascular resistance (SVR) by promoting the release of mediators such as serotonin, thromboxane A2, platelet-activating factor, and adenosine diphosphate. Serotonin is the most prominent mediator released. It is a potent pulmonary vasoconstrictor, and causes dilation of peripheral arterioles. Together, increased PVR in the presence of reduced RV preload causes a marked decrease in cardiac output (CO). Hypotension worsens as CO is increasingly affected (7). Ondansetron, a 5-hydroxytryptamine 3 (5-HT3) receptor antagonist, has been given preoperatively and intraoperatively to block serotonin-induced pulmonary vasoconstriction (7).

This study aimed to investigate whether blocking type 3 serotonin receptors with intravenous ondansetron would reduce hypotension due to bone cement syndrome in patients undergoing TKA under combined spinal-epidural anesthesia.

H0: Blocking type 3 serotonin receptors with intravenous ondansetron does not reduce hypotension due to bone cement syndrome.

H1: Blocking type 3 serotonin receptors with intravenous ondansetron reduces hypotension due to bone cement syndrome.

MATERIAL-METOD

This prospective randomized placebo-controlled, three-blind study will be conducted on patients aged ≥18 years, with unilateral TKA, ASA I-III physical condition, after obtaining informed written consent from The Atatürk University Medical Faculty Hospital ethics committee and patients. Patients with classical contraindications to subarachnoidal block, morbidly obese (body mass index > 35 kg / m2), hypersensitive to ondansetron and allergic to local anesthetic agents, taking selective serotonin reuptake inhibitors or serotonin-related migraine drugs, unstable angına, patients with hemodynamically severe aortic-mitral valve stenosis, severe carotid artery stenosis and severe pulmonary, renal, hepatic, cerebrovascular or psychiatric disease, neurological or cerebrovascular disease or psychiatric disease, hypertension but unable to take medication or arterial hypertension uncontrolled with oral medications, ASA>III, patients with preoperative anemia and patients who do not want to participate in the study will be excluded from the study. In all cases, antihypertensive drugs will be continued until the day of surgery.

The patients will be randomized by the statistician using a computerized random numbers table, with 12 individuals in each group, and divided into four equal groups. Group O (Ondansetron applied only, no tourniquet applied), Group TO (Ondansetron and tourniquet applied), Group S (No ondansetron and tourniquet applied), and Group TS (Ondansetron not applied, only tourniquet applied).

Ondansetron 0.15 mg/kg or 10 ml saline will be given intravenously 10 minutes before cement administration to the groups. At the same time, 100 ml of isolayt S will be administered together with the study drugs. Numbered opaque envelopes will be prepared in the order in which the randomization codes are. Corresponding authors and coauthors will evaluate patients' eligibility for the study, obtain informed consent, enroll patients, and analyze the collected data. The other investigator, blinded to the study groups, will perform spinal anesthesia, record intraoperative data, and give ıv drugs prepared by the primary investigator to the patient 10 minutes before cement administration. Neither patients, surgeons, nor people who evaluate patients intraoperatively and postoperatively will know what their study group is. Also, the study design will be three-blind, as the biostatistician who analyzes and interprets the data does not know what groups are.

A detailed anamnesis will be taken from the patients one day before the operation, a general system examination will be performed, and they will be informed about the study protocol and their written consent will be obtained. It will be stated to the patients that they should fast for 8 hours before the surgery and they can take clear liquids up to 2 hours before the surgery. When the patient comes to the operating room, two wide-lumen catheters (16-gauge) will be placed intravenously. After routine monitoring including electrocardiogram (ECG), pulse (NB), peripheral oxygen saturation (SpO2) and noninvasive blood pressure (NIBP), systolic arterial pressure (SAB), diastolic arterial pressure (DAP), mean arterial pressure (MAP), and also NB and Sp02 will be measured and these measurements will be recorded as baseline values. None of the patients will be sedated. The patients will be placed in a sitting position and combined spinal-epidural anesthesia will be applied from the midline. The skin will be sterilized. After infiltration of local anesthetic (2% lidocaine), an 18 gauge Tuohy needle will be advanced through the midline through the L2-3 or L3-4 intervertebral space. After the epidural space has been determined by the loss of resistance method, a 27 gauge pen-tipped needle will be inserted intrathecally using the needle-through-needle technique. After the free flow of cerebrospinal fluid is observed, 7.5 mg 0.5% isobaric bupivacaine and 15 µg fentanyl will be administered intrathecally within 30 seconds. The spinal needle will be removed and the epidural catheter will be fixed by placing 4-5 cm in the epidural space. The level of a sensory block will be evaluated by the loss of cold sensation, and surgery will be initiated when this level reaches T10-T12. If the block level is below T10, 5 ml of a solution containing 15 ml of 2% lidocaine + 2 ml of bicarbonate + 2 ml of fentanyl will be administered until the sensory block level above T10 is achieved through the epidural catheter. Patients will be given 15 mg/kg paracetamol and 50 mg dextoprufen as standard intraoperatively.

Motor block level will be evaluated with the modified Bromage scale. (0=patient can move hips, knees, ankles, and toes; 1=patient can fully flex foot and knee, unable to flex hip; 2=patient can flex the foot, unable to flex knee and hip; 3=total motor block).

Hemodynamic parameters and SpO2 will be recorded every 2 minutes for 20 minutes after combined spinal-epidural anesthesia, then every 5 minutes until bone cement is placed, every 2 minutes for 20 minutes after bone cement is placed, and then every 5 minutes until the end of the operation.

In the tourniquet group, these parameters were applied every 2 minutes for 20 minutes after combined spinal-epidural anesthesia, then every 5 minutes until the bone cement is placed, every 2 minutes for 20 minutes after the bone cement is placed, and every 5 minutes until the tourniquet is opened, after it is turned on every 2 minutes for 20 minutes and then every 5 minutes until the end of the operation.

At the end of the operation, the patients will be taken to the PACU, where hemodynamic parameters and SpO2 monitoring will continue to be recorded at 5-minute intervals.

Hypotension will be defined as a 20% decrease in systolic blood pressure from baseline. In this case, ephedrine, noradrenaline, and 200 ml of the rapid crystalloid or colloid solution will be administered. If bradycardia occurs (HR <50 beats/min) and bradycardia is not associated with hypotension, 1 mg of atropine IV will be given. If hypotension persists, inotropic drugs will be administered. Inotropic and vasopressor drugs will be administered according to the preference of the anesthesiologist. When the hematocrit drops to ≤30%, erythrocyte suspension will be given. The lowest systolic blood pressure recorded within 15 minutes of prosthesis insertion will be compared with the values 15 minutes before insertion, and in tourniquet users, the lowest systolic blood pressure recorded within 15 minutes after the tourniquet is deployed will be compared with the values 15 minutes before the tourniquet is deployed, and will be used to score the BCIS severity.

Sensory block levels of the patients will be recorded every 5 minutes intraoperatively.

Blood losses and necessary intraoperative fluids will be replaced before the cement is applied to the patients.

After the surgery, the patients will be evaluated in the recovery room. Visual analog scale (VAS; 0 cm = no pain, 10 cm = most severe pain), anesthesia-related side effects (eg, nausea or vomiting, and headache), and sensory block levels will be evaluated. If the patient's VAS is >3, 10 ml of 0.1% bupivacaine solution will be administered through the epidural catheter.

Patients' age, weight, height, BMI, gender, ASA, duration of operation, duration of anesthesia, preoperative hemoglobin, Bromage score, total doses of vasopressor, inotrope, atropine used, total amounts of blood, crystalloid and colloid used, comorbidities, drugs used, cement used amount, the highest level of sensory block, urinary output, duration of hypotension, number of patients who do not need vasopressors and inotropes, intraoperative nausea and vomiting, indication for surgery, tourniquet duration (Trauma, Arthrosis, Infectious, Necrosis Osteolysis) will be recorded.

If nausea and vomiting occur during the intraoperative period, metoclopramide (10 mg) will be given intravenously. QT prolongation, a side effect of study drugs, will be evaluated. QT prolongation will be defined as QT interval prolongation of more than half the previous RR interval on the ECG in the intraoperative and post-anesthetic care unit.

The primary outcome was hypotension occurring within 15 minutes after femoral bone cement placement.

The secondary outcome was hemodynamic changes, intraoperative sensory block level, nausea and vomiting, number of patients who did not need vasopressors, and inotropes during the operation.

POWER ANALYSIS

The SAP results in the reference article are given below (8). Considering SAP 158±20 before cementation and 20 minutes after cementation SAP 136±18.5, it was calculated with the G* power program that 12 patients should be included in the ondansetron group at 80% power at 95% confidence level.

In the design of the study, groups were determined as with and without ondansetron tourniquet, and with and without control tourniquet.

Therefore

* 12 patients who underwent ondansetron and tourniquet
* 12 patients without ondansetron and tourniquet
* 12 patients treated with saline (control) and tourniquet
* 12 patients without saline (control) and tourniquet A total of 48 patients were planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral TDA
* ASA I-III physical condition
* patients aged ≥18 years,

Exclusion Criteria:

* Patients with classical contraindications to subarachnoidal block,
* morbidly obese (body mass index > 35 kg / m2),
* hypersensitive to ondansetron and allergic to local anesthetic agents,
* taking selective serotonin reuptake inhibitors or serotonin-related migraine drugs,
* unstable angına,
* patients with hemodynamically severe aortic-mitral valve stenosis,
* severe carotid artery stenosis and severe pulmonary, renal, hepatic, cerebrovascular or psychiatric disease,
* neurological or cerebrovascular disease or psychiatric disease,
* hypertension but unable to take medication or arterial hypertension uncontrolled with oral medications,
* ASA>III physical condition,
* patients with preoperative anemia
* patients who do not want to participate in the study will be excluded from the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HYPOTENSION DUE TO BONE CEMENT SYNDROME IN TOTAL KNEE PROSTHESIS SURGERY
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Hypotension (mmHg) | Intraoperative
  The primary outcome was hypotension.Hypotension was defined as systolic blood pressure(mmHg) decrease exceeded 20% of baseline

SECONDARY OUTCOMES:
Systolic blood pressure (mmHg) | Intraoperative
  Change in systolic blood pressure (mmHg)
Diastolic blood pressure (mmHg) | Intraoperative
  Change in diastolic blood pressure (mmHg)
Heart rate (beats/min) | Intraoperative
  Change in heart rate (beats/min)

CONTACTS AND LOCATIONS:
Overall Officials: AYŞENUR DOSTBİL, Study Director — Ataturk University
Locations (1):
- Aysenur Dostbil, Yakutiye, Erzurum, Turkey (Türkiye)